CLINICAL TRIAL: NCT03740984
Title: Effects of Music or Hypnotherapy on Cancer Patients During Chemotherapy - A Prospective Off-centre Randomized Placebo-controlled Trial
Brief Title: Effects of Music or Hypnotherapy on Cancer Patients During Chemotherapy
Acronym: F-Chem
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn from sponsor.
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Collaborators: Deutsche Gesellschaft für hypnose und hypnotherapie E.V. (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Joscha Reinhard, Principal investigator, Dr. Horst Schmidt Klinik GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Gyn F-Chem
Record Dates: First submitted 2018-09-16; First posted 2018-11-14 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Breast Neoplasm; Ovary Cancer
Keywords: Chemotherapy; Side effects of chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective randomised Trial:
  Intervention 1 = hypnosis (hypnotherapy), Intervention 2 = Music therapy; Intervention 3 (Standard care)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Single blinded. The participant knows which group intervention is being used (music, hypnosis or standard care). This is being told while listening to the Intervention. All care Providers only know which "colour" mp3 player is being used (white, orange or black).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis / Hypnotherapy (Experimental): Hypnosis intervention has been created by a certified hypnosis therapist (Prof. Reinhard) has been audio-recorded. The hypnosis intervention is based on the patient's happy place as well as many other interventions which all focus on support and wellbeing (total recording time ca. 4 ½ hours). All patients are advice to start with the beginning, however during the course of chemotherapy they are allowed to skip mp3 files, if they prefer to listen to a new intervention.
  Interventions: Other: Interventions are self controlled by the patient via a mp3 player and noise reduction headphones.
- Music therapy (Experimental): For the music therapy the following music recordings have been used. All patients were allowed to skip tracks if they did not like to listen to that particular track.
  Purple Waves - Berlin Symphonic Film orchestra / Christopher Franke - Pacific Coast Highway Black Garden View - Berlin Symphonic Film orchestra / Christopher Franke - Pacific Coast Highway Sunset Destination - Berlin Symphonic Film orchestra / Christopher Franke - Pacific Coast Highway Crystal Tree - Berlin Symphonic Film orchestra / Christopher Franke - Pacific Coast Highway Best nature sounds / Ocean Volume 2 - Best Relaxation Music - Deep Sleep Top 10 Serse: Aria "Ombra mai Fu" - Andreas Scholl, Akademie für Alte music Berlin - Händel Johann Sebastian Bach: Jesus Bleibet Meine Freude (Studio) - Eduard Stan - Piano Recital Mozart: Concerto pour violon no 4 en re majeur, KV (Köchel listing) 218 - Christian Ferras; Pietro Argento; Orchestra Scarlatti di Nap - La fete a Stradivarius
  ... etc.
  Interventions: Other: Interventions are self controlled by the patient via a mp3 player and noise reduction headphones.
- Standard therapy (Placebo Comparator): In this standard therapy the patient listens to a short explanation that they were randomized into the control arm and that they are allowed to listen to silence (tracks with no music or intervention).
  Interventions: Other: Interventions are self controlled by the patient via a mp3 player and noise reduction headphones.

INTERVENTIONS:
Other: Interventions are self controlled by the patient via a mp3 player and noise reduction headphones. — During premedication and during chemotherapy the patient is connected to a long term ECG recording and allowed to listen to the mp3 Player via noise reduction headphones.

SUMMARY:
Chemotherapies often induce side effects. This study examines whether hypnosis, music therapy versus standard therapy influence these side effects.

DETAILED DESCRIPTION:
Primary study goals are differences in quality of life, nausea and vomiting episodes, fatigue, depression and change of taste.

ELIGIBILITY:
Inclusion Criteria:

* no previous chemotherapy
* compliance of the patient to fill out questionnaires
* informed consent and signed forms
* histologic secured breast cancer or ovary cancer (residual tumor after surgery equal or less than 0,5 cm)
* One of following chemotherapy regime:

  4x Epirubicin / Cyclophosphamid, 12x paclitaxel oder 6x Carboplatin / Docetaxel / Perjeta/ Herceptin oder 6x Doxorubicin, docetaxel, Cyclophosphamid oder 6 x Carboplatin / paclitaxel + / - Avastin oder 4x Epirubicin / Cyclophosphamid -> 12x paclitaxel /herceptin/ perjeta oder 4x Epirubicin / Cyclophosphamid q21->12xcarboplatin, paclitaxel 4 Epirubicin / Cyclophosphamid q14-> 12 carboplatin, paclitaxel

Exclusion Criteria:

* does not understand the German language
* psychosis
* not able to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
ZSDS = Zung Self-rating Depression Scale | Every three weeks during chemotherapy and one year after last chemotherapy
  Change of questionnaire scores
Quality of life questionnaire - Core30 | Every three weeks during chemotherapy and one year after last chemotherapy
  Change of questionnaire scores
Patient diary, number of emetic episodes, the intensity of Nausea and QoL evaluation (functional living index-emesis questionnaire) | Day 1-5 after chemotherapie and before next chemotherapy
  Change of questionnaire scores
Fatigue assessment questionnaire (FAQ) | Every three weeks during chemotherapy and one year after last chemotherapy
  Change of questionnaire scores
Screening Scale for Taste Alteration (TA) | Every three weeks during chemotherapy and one year after last chemotherapy
  Change of questionnaire scores

SECONDARY OUTCOMES:
Change of heart rate | change of average heart rate after 5 minutes rest, 5 minutes before chemotherapy and 5 minutes into chemotherapy
  Long term ECG recording before and during chemotherapy

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Klinik für Gynäkologie und gynäkologischen Onkologie, Wiesbaden, Hesse
  - Helios Berlin Buch, Berlin
  - Helios Kliniken Schwerin GmbH, Schwerin

IPD SHARING:
Plan to Share IPD: No